CLINICAL TRIAL: NCT01696058
Title: A Randomised, Double Blind, Parallel Group Study to Assess the Efficacy and Safety of 12 Weeks of Once Daily, Orally Inhaled, Co-administration of Olodaterol 5µg (Delivered by the Respimat® Inhaler) and Tiotropium 18µg (Delivered by the HandiHaler®) Compared to Once Daily, Orally Inhaled, Co-administration of Placebo (Delivered by the Respimat® Inhaler) and Tiotropium 18µg (Delivered by the HandiHaler®) in Patients With Chronic Obstructive Pulmonary Disease (COPD)[ANHELTO TM 2]
Brief Title: Co-administration of Olodaterol Respimat® and Tiotropium Handihaler®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.52
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

ARMS (2):
- Olodaterol andTiotropium (Experimental): 2 puffs Olodaterol from Respimat and one capsule Tiotropium by Handihaler once daily in am, co-administered
  Interventions: Drug: Tiotropium; Drug: Olodaterol
- Placebo and Tiotropium (Other): 2 puffs placebo inhalation solution from Respimat and one capsule Tiotropium by Handihaler once daily in am, co-administered
  Interventions: Drug: Tiotropium; Drug: Placebo matching Olodaterol

INTERVENTIONS:
Drug: Tiotropium — marketed product
  Arms: Placebo and Tiotropium
Drug: Placebo matching Olodaterol — one dose
  Arms: Placebo and Tiotropium
Drug: Tiotropium — marketed product
  Arms: Olodaterol andTiotropium
Drug: Olodaterol — one dose
  Arms: Olodaterol andTiotropium

SUMMARY:
The overall objective of this study is to assess efficacy and safety of 12 weeks, once daily, orally inhaled co-administration of olodaterol 5 µg (delivered by the Respimat® Inhaler) and tiotropium (delivered by the Handihaler® as Spiriva Handihaler®), compared to tiotropium (Spiriva Handihaler®) monotherapy on lung function in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria: Patients must have a relatively stable airway obstruction with a post-bronchodilator FEV1 ≥ 30 % and < 80% of predicted normal and a post-bronchodilator FEV1/FVC <70% at Visit 1.
3. Male or female patients, 40 years of age or older.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to: perform technically acceptable pulmonary function tests, and maintain records(paper diary).
6. Patients must be able to inhale medication in a competent manner from the Respimat Inhaler as well as the Handihaler.

Exclusion criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patients ability to participate in the study.
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an AST >x2 ULN, ALT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN will be excluded regardless of clinical condition (a repeat laboratory evaluation will not be conducted in these patients).
3. Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma. If a patient has a total blood eosinophil count ≥600/mm3, source documentation is required to verify that the increased eosinophil count is related to a non-asthmatic condition.
4. A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists).
5. A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists).
6. A history of myocardial infarction within 1 year of screening visit (Visit 1).
7. Unstable or life-threatening cardiac arrhythmia.
8. Hospitalization for heart failure within the past year.
9. Known active tuberculosis.
10. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed).
11. A history of life-threatening pulmonary obstruction.
12. A history of cystic fibrosis.
13. Clinically evident bronchiectasis.
14. A history of significant alcohol or drug abuse.
15. Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1).
16. Patients being treated with oral or patch ß-adrenergics.
17. Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
18. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigators opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
19. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program.
20. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit (Visit 1).
21. Patients with known hypersensitivity to ß-adrenergic drugs, BAC, EDTA, or any other component of the Respimat® inhalation solution.
22. Patients with known hypersensitivity to anticholinergic drugs, lactose, or any other components of the HandiHaler®.
23. Pregnant or nursing women.
24. Women of childbearing potential not using a highly effective method of birth control*. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.

    * as per ICH M3(R2) a highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year).
25. Patients who have previously been randomised in this study or are currently participating in another study.
26. Patients who are unable to comply with pulmonary medication restrictions prior to randomisation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1137 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (94):
- United States (94):
  - 1222.52.02090 Boehringer Ingelheim Investigational Site, Anniston, Alabama
  - 1222.52.02046 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1222.52.02014 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1222.52.02017 Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - 1222.52.02092 Boehringer Ingelheim Investigational Site, Anchorage, Alaska
  - 1222.52.02072 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1222.52.02063 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1222.52.02088 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 1222.52.02012 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1222.52.02006 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1222.52.02031 Boehringer Ingelheim Investigational Site, San Jose, California
  - 1222.52.02011 Boehringer Ingelheim Investigational Site, Torrance, California
  - 1222.52.02061 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1222.52.02054 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1222.52.02001 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1222.52.02037 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1222.52.02055 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1222.52.02094 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.52.02022 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1222.52.02074 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1222.52.02016 Boehringer Ingelheim Investigational Site, Ponte Verda, Florida
  - 1222.52.02084 Boehringer Ingelheim Investigational Site, Saint Petersberg, Florida
  - 1222.52.02043 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1222.52.02009 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1222.52.02048 Boehringer Ingelheim Investigational Site, Duluth, Georgia
  - 1222.52.02077 Boehringer Ingelheim Investigational Site, Gainsville, Georgia
  - 1222.52.02040 Boehringer Ingelheim Investigational Site, Rincon, Georgia
  - 1222.52.02024 Boehringer Ingelheim Investigational Site, O'Fallon, Illinois
  - 1222.52.02002 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 1222.52.02008 Boehringer Ingelheim Investigational Site, Fort Mitchell, Kentucky
  - 1222.52.02025 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1222.52.02089 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1222.52.02005 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1222.52.02029 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1222.52.02036 Boehringer Ingelheim Investigational Site, Hollywood, Maryland
  - 1222.52.02015 Boehringer Ingelheim Investigational Site, Townson, Maryland
  - 1222.52.02034 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1222.52.02003 Boehringer Ingelheim Investigational Site, Chelsea, Michigan
  - 1222.52.02020 Boehringer Ingelheim Investigational Site, Kalamazoo, Michigan
  - 1222.52.02047 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1222.52.02049 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1222.52.02079 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 1222.52.02068 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 1222.52.02028 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1222.52.02053 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1222.52.02050 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 1222.52.02035 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1222.52.02030 Boehringer Ingelheim Investigational Site, Marlton, New Jersey
  - 1222.52.02071 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1222.52.02064 Boehringer Ingelheim Investigational Site, Johnson City, New York
  - 1222.52.02087 Boehringer Ingelheim Investigational Site, New Windsor, New York
  - 1222.52.02091 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 1222.52.02076 Boehringer Ingelheim Investigational Site, Calabash, North Carolina
  - 1222.52.02010 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1222.52.02045 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1222.52.02038 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1222.52.02051 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1222.52.02058 Boehringer Ingelheim Investigational Site, Tabor City, North Carolina
  - 1222.52.02013 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1222.52.02062 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1222.52.02039 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1222.52.02081 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1222.52.02093 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1222.52.02059 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1222.52.02026 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1222.52.02097 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1222.52.02075 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1222.52.02102 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1222.52.02080 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1222.52.02100 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1222.52.02096 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1222.52.02085 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.52.02101 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.52.02065 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 1222.52.02042 Boehringer Ingelheim Investigational Site, Myrtle Beach, South Carolina
  - 1222.52.02083 Boehringer Ingelheim Investigational Site, Rock Hill, South Carolina
  - 1222.52.02066 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.52.02095 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.52.02098 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1222.52.02018 Boehringer Ingelheim Investigational Site, Brentwood, Tennessee
  - 1222.52.02086 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1222.52.02044 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1222.52.02041 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 1222.52.02027 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1222.52.02056 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1222.52.02007 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1222.52.02060 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1222.52.02078 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
  - 1222.52.02082 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1222.52.02057 Boehringer Ingelheim Investigational Site, Midvale, Utah
  - 1222.52.02023 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.52.02069 Boehringer Ingelheim Investigational Site, Selah, Washington
  - 1222.52.02019 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1222.52.02099 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] ZuWallack R, Allen L, Hernandez G, Ting N, Abrahams R. Efficacy and safety of combining olodaterol Respimat((R)) and tiotropium HandiHaler((R)) in patients with COPD: results of two randomized, double-blind, active-controlled studies. Int J Chron Obstruct Pulmon Dis. 2014 Oct 14;9:1133-44. doi: 10.2147/COPD.S72482. eCollection 2014. PMID 25342898

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1137 patients were entered and randomized to treatment and 1135 patients were treated with study medication.
Groups:
- Olodaterol (5μg) and Tiotropium (18μg): 2 puffs olodaterol from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Olodaterol: One dose
  Tiotropium: Marketed dose
- Placebo and Tiotropium (18μg): 2 puffs placebo inhalation solution from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Tiotropium: Marketed dose, 2 inhalations from 1 capsule once daily in the morning
  Placebo matching Olodaterol: One dose, 2 inhalations once daily in the morning
Period: Overall Study
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Started | 566 | 569
Completed | 523 | 538
Not Completed | 43 | 31
Not completed — Adverse Event | 21 | 11
Not completed — Lack of Efficacy | 2 | 3
Not completed — Protocol Violation | 9 | 3
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Other reason prematurely discontinued | 5 | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS), which includes all randomized patients who receive at least one dose of double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg) | Total
Number analyzed (Participants) | 566 | 569 | 1135
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.0) | 63.6 (8.9) | 64.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 261 | 266 | 527
  Male | 305 | 303 | 608

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-3h Response at 12 Weeks; Defined as Change From Baseline to Week 12
Description: FEV1 (Forced expiratory volume in 1 second) AUC0-3h (area under the curve) response at 12 weeks; defined as change from baseline to Week 12. AUC was standardized by dividing by time unit.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks. FAS included all patients in the treated set who had both baseline and at least one post-baseline measurement at or before 12 weeks for any of the co-primary efficacy variables
Measure: Least Squares Mean (Standard Error); unit: Area Under the Curve (L) (standardized)
Groups:
- Olodaterol (5μg) and Tiotropium (18μg): 2 puffs olodaterol from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Olodaterol: One dose, 2 inhalations once daily in the morning
  Tiotropium: Marketed dose, 2 inhalations from 1 capsule once daily in the morning
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 563 | 566
Area Under the Curve (L) (standardized) | 0.297 (0.010) | 0.191 (0.010)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Results are from an mixed model repeated measure (MMRM) model. Fixed effects include treatment, visit, treatment by visit interaction, baseline and baseline by visit interaction. Patient is considered random and an unstructured covariance structure was used. Number of patients contributing to models: Tio+Placebo (566), Tio+Olo 5ug (563); Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.078 to 0.135], Standard Error of Mean 0.014

2. Primary Outcome: Trough FEV1 Response at 12 Weeks; Defined as Change From Baseline to Week 12
Description: Trough FEV1 (Forced expiratory volume in 1 second) response at 12 weeks; defined as change from baseline to Week 12
Time Frame: baseline and 12 weeks
Population: Full Analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 550 | 555
L | 0.175 (0.009) | 0.135 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Results are from an MMRM model. Fixed effects include treatment, visit, treatment by visit interaction, baseline and baseline by visit interaction. Patient is considered random and an unstructured covariance structure was used. Number of patients contributing to models: Tio+Placebo (555), Tio+Olo 5ug (550); Test type: Superiority or Other; p = 0.0029, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [0.014 to 0.065], Standard Error of Mean 0.013

3. Secondary Outcome: Saint George Respiratory Questionnaire - (Total Score) Based on Combined 1222.51 and 1222.52 Data
Description: The Saint George Respiratory Questionnaire (SGRQ) is designed to measure health impairment in patients with asthma and chronic obstructive pulmonary disease (COPD). It is divided into two parts. Part I produces the Symptoms score (several scales), and Part II the Activity and Impacts scores [dichotomous (true/false) except last question (4-point Likert scale)]. A Total score is also produced with scores ranging from 0 to 100, with higher scores indicating more limitations. Since the SGRQ analysis is based on the combined data from both this study and protocol 1222.51 (NCT01694771), only combined SGRQ results will be included in the latest clinical trial report. Hence there will only be one SGRQ analysis from both studies, which will not appear in the first clinical trial report. For this same reason, another covariate - study - will also be included in the MMRM for SGRQ analysis. The combined data for this outcome measure was pre-specified in both protocols.
Time Frame: 12 weeks
Population: FAS with last observation carried forward (LOCF) imputation (combined data from twin studies 1222.51 and 1222.52). Number of patients contributing to models: Tio+Placebo (1055), Tio+Olo 5ug (1039).
Measure: Least Squares Mean (Standard Error); unit: units on a scale (total score)
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 1039 | 1055
units on a scale (total score) | 41.204 (0.327) | 43.059 (0.325)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Results are from ANCOVA model. Fixed effects include study, treatment and baseline. Number of patients contributing to models: Tio+Placebo (1055), Tio+Olo 5ug (1039); Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.854, 95% CI 2-sided [-2.757 to -0.951], Standard Error of Mean 0.461

4. Secondary Outcome: Peak FEV1 Response at 12 Weeks - Defined as Change From Baseline
Description: Peak FEV1 (Forced Expiratory Volume in 1 second) response at 12 Weeks - defined as change from baseline. All p-values for these measures are only descriptive.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 563 | 566
L | 0.371 (0.011) | 0.271 (0.011)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Results are from an MMRM model. Fixed effects include treatment, visit, treatment by visit interaction, baseline and baseline by visit interaction. Patient is considered random and an unstructured covariance structure was used. Number of patients contributing to models: Tio+Placebo (566), Tio+Olo 5ug (563); Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [0.071 to 0.129], Standard Error of Mean 0.015

5. Secondary Outcome: FVC AUC0-3h Response at 12 Weeks; Defined as Change From Baseline
Description: Forced Vital Capacity (FVC) AUC0-3h response at 12 weeks - defined as change from baseline. AUC was standardized by dividing by time unit.
Time Frame: baseline and 12 Weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 563 | 566
L | 0.424 (0.017) | 0.306 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [0.072 to 0.164], Standard Error of Mean 0.023

6. Secondary Outcome: Peak FVC Response at 12 Weeks; Defined as Change From Baseline
Description: Peak FVC response at 12 weeks - defined as change from baseline.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 563 | 566
L | 0.562 (0.017) | 0.457 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [0.057 to 0.152], Standard Error of Mean 0.024

7. Secondary Outcome: Trough FVC Response at 12 Weeks; Defined as Change From Baseline
Description: Trough Forced Vital Capacity (FVC) response at 12 weeks- defined as change from baseline.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 550 | 555
L | 0.269 (0.015) | 0.235 (0.015)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1156, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.008 to 0.076], Standard Error of Mean 0.022

8. Secondary Outcome: Rescue Medication Usage - Percentage of Rescue Free Days
Description: Rescue medication usage - the percentage of rescue free days. The percentage of rescue free days is defined as: number of rescue free days divided by total exposure, multiplied by 100%. The baseline for the number of rescue-free days was defined as the number of rescue-free days observed during the last week of the baseline period (i.e., the 7 days prior to administration of the first dose of randomized treatment).
  Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline.
  Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (552)
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 552 | 559
percentage of days
  Week 1 | 53.207 (1.481) | 48.583 (1.472)
  Week 2 | 54.249 (48.640) | 48.640 (1.477)
  Week 3 | 54.820 (1.536) | 49.865 (1.528)
  Week 4 | 60.761 (1.388) | 55.969 (1.378)
  Week 5 | 60.154 (1.550) | 51.840 (1.549)
  Week 6 | 59.707 (1.572) | 49.001 (1.568)
  Week 7 | 59.493 (1.598) | 50.164 (1.594)
  Week 8 | 59.021 (1.634) | 51.017 (1.626)
  Week 9 | 60.524 (1.636) | 51.273 (1.620)
  Week 10 | 60.216 (1.636) | 51.634 (1.616)
  Week 11 | 59.650 (1.636) | 51.604 (1.616)
  Week 12 | 62.327 (1.525) | 55.090 (1.508)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Week 12: Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline. Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (552); Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean difference from Tio+Placebo Week 12 = 7.237, 95% CI 2-sided [3.028 to 11.446], Standard Error of Mean 2.145

9. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Total Daily)
Description: Rescue medication usage - mean weekly rescue usage (total daily). The baseline for the rescue use was the mean of the observations during the last week of the baseline period. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol metered dose inhaler (MDI) (100 μg per puff) was provided as rescue medication . Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
  Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline.
  Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (555)
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: usage (total daily) number of puffs
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 555 | 559
usage (total daily) number of puffs
  Week 1 | 1.627 (0.066) | 2.072 (0.066)
  Week 2 | 1.652 (0.072) | 2.145 (0.072)
  Week 3 | 1.635 (0.078) | 2.167 (0.078)
  Week 4 | 1.647 (0.081) | 2.189 (0.080)
  Week 5 | 1.551 (0.081) | 2.183 (0.080)
  Week 6 | 1.523 (0.081) | 2.179 (0.080)
  Week 7 | 1.540 (0.083) | 2.138 (0.082)
  Week 8 | 1.586 (0.085) | 2.107 (0.084)
  Week 9 | 1.519 (0.083) | 2.121 (0.082)
  Week 10 | 1.499 (0.082) | 2.103 (0.081)
  Week 11 | 1.484 (0.083) | 2.107 (0.082)
  Week 12 | 1.535 (0.084) | 2.103 (0.083)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); Week 12 - Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline. Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (555); Test type: Superiority or Other; p < .0001, ANCOVA; Mean difference from Tio+Placebo Week 12 = -0.568, 95% CI 2-sided [-0.800 to -0.336], Standard Error of Mean 0.118

10. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Daytime)
Description: Rescue medication usage - Mean weekly rescue usage during daytime hours. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol MDI (100 μg per puff) was provided as rescue medication by BI, and only the albuterol MDI provided by BI was allowed for rescue medication use. Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
  Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline.
  Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (555)
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 555 | 559
number of puffs
  Week 1 | 0.406 (0.025) | 0.437 (0.025)
  Week 2 | 0.421 (0.027) | 0.466 (0.027)
  Week 3 | 0.407 (0.030) | 0.459 (0.030)
  Week 4 | 0.408 (0.031) | 0.479 (0.031)
  Week 5 | 0.375 (0.030) | 0.479 (0.030)
  Week 6 | 0.378 (0.030) | 0.491 (0.030)
  Week 7 | 0.403 (0.033) | 0.499 (0.032)
  Week 8 | 0.417 (0.033) | 0.482 (0.033)
  Week 9 | 0.396 (0.033) | 0.487 (0.032)
  Week 10 | 0.392 (0.032) | 0.480 (0.031)
  Week 11 | 0.383 (0.031) | 0.482 (0.031)
  Week 12 | 0.393 (0.032) | 0.483 (0.032)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0467, ANCOVA; Mean difference from Tio+Placebo Week 1 = -0.090, 95% CI 2-sided [-0.178 to -0.001], Standard Error of Mean 0.045

11. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Nighttime)
Description: Rescue medication usage - Mean weekly rescue usage during nighttime hours. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol MDI (100 μg per puff) was provided as rescue medication by BI, and only the albuterol MDI provided by BI was allowed for rescue medication use. Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
  Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline.
  Number of patients contributing to models: Tio+Placebo (559), Tio+Olo 5ug (555)
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Number analyzed (Participants) | 555 | 559
number of puffs
  Week 1 | 1.222 (0.055) | 1.633 (0.055)
  Week 2 | 1.232 (0.058) | 1.677 (0.058)
  Week 3 | 1.229 (0.062) | 1.707 (0.062)
  Week 4 | 1.239 (0.064) | 1.709 (0.064)
  Week 5 | 1.177 (0.065) | 1.710 (0.064)
  Week 6 | 1.148 (0.065) | 1.692 (0.064)
  Week 7 | 1.139 (0.065) | 1.641 (0.064)
  Week 8 | 1.173 (0.067) | 1.628 (0.066)
  Week 9 | 1.125 (0.065) | 1.636 (0.065)
  Week 10 | 1.108 (0.066) | 1.630 (0.065)
  Week 11 | 1.104 (0.067) | 1.630 (0.066)
  Week 12 | 1.143 (0.067) | 1.625 (0.066)
Statistical Analysis 1: Comparison: Olodaterol (5μg) and Tiotropium (18μg) vs Placebo and Tiotropium (18μg); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; Mean difference from Tio+Placebo Week 12 = -0.483, 95% CI 2-sided [-0.668 to -0.298], Standard Error of Mean 0.094

ADVERSE EVENTS:
Time Frame: Adverse events were to be documented throughout the trial, i.e., starting with informed consent and ending 21 days after last administration of trial medication. the duration of treatment was up to 12 weeks.
Arm/Group | Olodaterol (5μg) and Tiotropium (18μg) | Placebo and Tiotropium (18μg)
Serious Adverse Events (participants affected / at risk) | 24/566 | 27/569
Other Adverse Events (participants affected / at risk) | 48/566 | 44/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5μg) and Tiotropium (18μg) (N=566) | Placebo and Tiotropium (18μg) (N=569)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5μg) and Tiotropium (18μg) (N=566) | Placebo and Tiotropium (18μg) (N=569)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 48 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.